CLINICAL TRIAL: NCT06225050
Title: A Single-center Pilot Study Using TCRα/β and CD45RA Depleted Stem Cell Grafts From Haploidentical Donors for Hematopoietic Cell Transplantation in Adults(HAPLO2022)
Brief Title: M-2018-334 in Hematological Malignancies
Acronym: HAPLO2022
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Collaborators: City of Hope Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-2018-334
Record Dates: First submitted 2023-12-05; First posted 2024-01-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- HSC Recipient (Experimental): PBSC grafts from haploidentical donors depleted of TCRaβ+ cells and CD45RA+ cells using CliniMACS Prodigy® will be infused into patients intravenously (IV)
  Interventions: Device: CliniMACS Prodigy® LP-TCRα/β-19-45RA (Trial Version)

INTERVENTIONS:
Device: CliniMACS Prodigy® LP-TCRα/β-19-45RA (Trial Version) — PBSC grafts from haploidentical donors depleted of TCRaβ+ cells and CD45RA+ cells using CliniMACS Prodigy® will be infused into patients intravenously (IV)

SUMMARY:
This is a single-center, open-label, single-arm, pilot clinical study using TCRα/β and CD45RA depleted stem cell grafts from haploidentical donors for hematopoietic cell transplantation in 12 to 18 adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients, between 18 years to 75 years of age, with high-risk hematological malignancy requiring an allogeneic hematopoietic stem cell transplantation (AlloHCT), but do not have an HLA-matched donor available

Exclusion Criteria:

* <3 months after preceding autologous transplantation or prior AlloHCT
* History of neurological impairment (active seizures, severe peripheral neuropathy, signs of leukoencephalopathy, active CNS infection)
* Active fungal infections with radiological and clinical progression
* Liver function abnormalities with bilirubin >2 mg/dL and elevation of transaminases higher than 400 U/L
* Chronic active viral hepatitis
* Cardiac dysfunction: adult patients ejection fraction <50% on echocardiography
* Patients with uncontrolled, >grade II hypertension (per Common Toxicity Criteria, CTC)
* Creatinine clearance <60 mL/min/1.73m2
* Respiratory failure necessitating supplemental oxygen
* HIV infection
* Positive anti-donor HLA antibody
* Treatment with checkpoint inhibitors in the period between 3 months prior to and 3 months after transplantation
* Female patients who are pregnant or breast feeding, or adults of reproductive potential not willing to use an effective method of birth control during study treatment and for at least 12 months thereafter. Note: Women of childbearing potential must have a negative serum pregnancy test at study entry
* Concurrent severe or uncontrolled medical disease (e.g., uncontrolled diabetes, myocardial infarction within 6 months prior to the study) which by assessment of the treating physician could compromise participation in the study
* Patients with a history of psychiatric illness or a condition which could interfere with their ability to understand the requirements of the study (this includes alcoholism/drug addiction).
* Patients unwilling or unable to comply with the protocol or unable to give informed consent
* Treatment with any investigational product within 4 weeks prior to study treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe acute GVHD (aGVHD) till Day 100 | 100 days after haploidentical hematopoietic cell transplantation
  Participants will be evaluated for the occurrence of aGVHD, grades III-IV in the first 100 days after transplantation and the time to occurrence of aGVHD, grades III-IV will be recorded. Severity of acute GVHD will be graded according to the CONSENSUS CRITERIA FOR GRADING OF ACUTE GVHD which has four Grades from Grade I to Grade IV. The higher the Score, the Worse the outcome.

SECONDARY OUTCOMES:
Performance of the CliniMACS Prodigy® LP-TCRα/β-19-45RA(Trial Version) | Until Last Patient Last Visit(24 Months)
  Performance of the CliniMACS Prodigy® LP-TCRα/β-19-45RA (Trial Version) will be assessed by calculating the log-depletion of TCRα/β+ and CD45RA+ cells
Incidence of acute GVHD (aGVHD) till six months post-transplantation | 6 Months
  Incidence of aGVHD, grade II-IV till six months post-transplantation will be evaluated. The maximum grade and the time to occurrence of acute GVHD will be recorded. Incidence and severity of acute GVHD will be graded according to the Consensus Criteria
Neutrophil Engraftment | Day 7
  Time to neutrophil engraftment will be defined as the first of three consecutive measurements of ANC ≥500/µL following conditioning regimen induced nadir, starting from the day of the first stem cell transplantation
Platelet Engraftment | Day 0
  Time to platelet engraftment will be defined as the first of three consecutive measurements of platelet count ≥20,000/µL without platelet transfusion support, starting from the day of the first stem cell transplantation.
Chronic GVHD | 1 Year
  Incidence and severity of chronic GVHD will be graded according to standard criteria for grading of chronic GVHD
Non-relapse mortality (NRM) | Until Last patient last Visit(24 Months)
  NRM is defined as death occurring in a patient between the first day of conditioning and day of last assessment (all visits throughout the study), not due to disease relapse/recurrence
Infusion toxicity | 15 minutes, 30 minutes, 2 hours, and 4 hours post infusion
  Maximum infusion toxicity on the days of transfusion will be evaluated by measuring the patient's blood pressure, heart rate, respiration rate and temperature one hour prior to the allograft infusion and then approximately 15 minutes, 30 minutes, 2 hours, and 4 hours post infusion
Graft failure | 30 Days
  Primary graft failure is defined as the failure to achieve an ANC ≥500 cells/µL by Day +30 in the setting of donor chimerism < 5% using local methods
Overall survival (OS) | Day 100 and through study completion, an average of 1 year post transplantation
  OS defined as time from transplantation to death or last follow-up and will be assessed at Day 100 and after 1 year
Disease-free survival (DFS) | Day 100 and through study completion, an average of 1 year post transplantation
  DFS is defined as the minimum time to relapse/recurrence, to death or to the last follow-up, from the time of transplantation and will be assessed at Day 100 and after 1 year
GVHD/relapse-free survival (GRFS) | GRFS will be assessed at Month 12 post transplantation
  An event is defined as grade III-IV acute GVHD, moderate to severe chronic GVHD, disease relapse, or death by any cause. GRFS will be assessed at 1 year.
Immunosuppression-free survival (ISFS) | Assessed at 1 year with a starting point at Day 45 post-transplantation
  Defined as being alive, relapse-free and off immunosuppressive therapy and will be assessed at 1 year with a starting point at Day 45 post-transplantation. Immune suppression is defined as any systemic agents used to control or suppress GVHD.
Relapse rate | 12 Months
  Time to relapse will be calculated from the time of transplantation to evidence of relapse
Hospitalization length/re-admission | Assessed at Day 30, Day 100 and at 12 Months post transplantation
  Number of days that patients had to be hospitalized until discharge after transplantation, and after any subsequent occurrence of an event leading to re- hospitalization assessed

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A multi-center phase I/II safety and feasibility study using CliniMACS TCRα/β and CD19 depleted stem cell grafts from haploidentical donors for hematopoietic progenitor cell transplantation in children and adults" — https://www.clinicaltrialsregister.eu/ctr-search/trial/2011-005562-38/results